CLINICAL TRIAL: NCT00365742
Title: Simvastatin Vs Therapeutic Lifestyle Changes and Supplements: A Primary Prevention Randomized Trial
Brief Title: Statin Therapy Vs. Therapeutic Lifestyle Changes and Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Hill Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWA00005390-Chestnut Hill Hosp
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2006-08-17 (Estimated); Status verified 2006-08

CONDITIONS: Hyperlipidemia
Keywords: red yeast rice; pharmaceutical grade fish oil; simvastatin; primary prevention
MeSH Terms: conditions — Hyperlipidemias | interventions — Simvastatin; red yeast rice

INTERVENTIONS:
Drug: simvastatin
Drug: red yeast rice
Drug: pharmaceutical grade fish oil
Behavioral: therapeutic lifestyle changes

SUMMARY:
Randomized trial in a primary prevention population

* all participants have high LDL cholesterol

Group one will take simvastatin 40 mg/day Group Two will make therapeutic lifestyle changes,and take supplements consisting of red yeast rice and fish oil

DETAILED DESCRIPTION:
This is a randomized primary prevention trial to compare the LDL lowering effects of an alternative regimen to statins(simvastatin) This alternative regimen is over the counter and available at health food stores. The alternative regimen consists of lifestyle changes including a Mediterranean Diet,exercise program, and stress reduction, with red yeast rice 1200 mg twice per day and fish oil 6 grams/day. The second group, run at the same time will take Zocor(simvastatin) 40 mg per day with standard counseling

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-75 yrs, who meet ATP III criteria to be treated for high cholesterol. All participants must be able to exercise and be willing to be randomized to either arm of the study

Exclusion Criteria:

* No history of bypass surgery, stents, or hx of myocardial infarction. Cannot have uncontrolled hypertension(SBP>190 or DBP>100), cannot have known intolerance to one of the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-04; Study Completion 2006-06

PRIMARY OUTCOMES:
LDL-c cholesterol

SECONDARY OUTCOMES:
total cholesterol
HDL
Triglycerides
cardiac CRP

CONTACTS AND LOCATIONS:
Overall Officials: David Becker, Principal Investigator